CLINICAL TRIAL: NCT04510961
Title: Beneficial Effects of Paraffin Bath Therapy as Additional Treatment of Chronic Hand Eczema: A Randomized Controlled Trial
Brief Title: Paraffin Bath Therapy for Chronic Hand Eczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ZIZI MOHAMMED IBRAHIM ALI, ASSOCIATE PROF, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Paraffin Hand Eczema
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Eczema
Keywords: Paraffin bath therapy, Hand Eczema, SCORAD, DLQI, Itching
MeSH Terms: conditions — Eczema; Pruritus

STUDY DESIGN:
Intervention Model Description: Sixty patients with moderate to severe Chronic Hand eczema (CHE) will participate in the study. They will be classified randomly into two groups of equal number; paraffin group and the control group.
  Interventions: Paraffin group will receive Paraffin Therapy for 5 days per week for 12 weeks in addition to routine skin care program while the control group will received routine skin care program
Who Masked: Outcomes Assessor
Masking Description: Measurements will be at three occasions: at randomization (T1), at 6th week (T2) and at 12th week (T3) of treatment. Evaluative procedures will be by a blind assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paraffin baths therapy (PBT) :group A (Active Comparator): Patients in treatment group will receive paraffin wax baths for five days per week for 12 weeks.
  Interventions: Other: Paraffin baths therapy
- Control group (B) (No Intervention): receive routine skin care program ; lifestyle change, emollients and moisturizers

INTERVENTIONS:
Other: Paraffin baths therapy — Patients in treatment group will receive paraffin wax baths for five days per week for 12 weeks. Prepare the paraffin device and blocks of paraffin wax. Put the paraffin wax blocks inside the tank and set the thermostat 35 to 40◦C. Melting paraffin was taken from 90 to 120 minutes. Adjust the suitable temperature for each patient before immersion of patient's hand. Submerge patient's hand completely for three to four seconds then withdraw it
  Arms: Paraffin baths therapy (PBT) :group A

SUMMARY:
Objective: Chronic Hand eczema (CHE) is a common inflammatory skin disease has a major medical psychological and socio-economic implications that affect quality of life (QoL)and work ability. This study, the first randomized controlled trial that will be conducted to evaluate the effect of paraffin bath therapy (PBT) in the treatment of CHE.

DETAILED DESCRIPTION:
Design: The study design is a randomized controlled trial with measures at pre-and post-intervention.

Subjects: Sixty patients with moderate to severe Chronic Hand eczema (CHE) will participate in the study. They will be classified randomly into two groups of equal number; paraffin group and the control group.

Interventions: Paraffin group will receive Paraffin bath therapy for 5 days per week for 12 weeks in addition to routine skin care program while the control group will receive routine skin care program.

Outcome Measures:

Objective SCORing Atopic Dermatitis, subjective item score and dermatology life quality index (DLQI) will be assessed before, at 6th week and at 12th week of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20-40 years
* Time elapsed from the beginning of the disease ; more than three months according to the Guideline of the German Dermatological Society

Exclusion Criteria:

* active eczematous lesions on other parts of the body;
* malignant or premalignant skin tumors

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
SCORAD ("SCORing Atopic Dermatitis | Change from Baseline at SCORAD score at 6th week and at 12th weeks of treatment
  is the most widely clinical tool for assessing the severity (i.e. extent, intensity) of atopic dermatitis as objectively as possible.20 It consists of six objective items (erythema, oedema/papules, effect of scratching, oozing/crust formation, lichenification, and dryness), and two subjective symptoms (itch and sleeplessness), the maximum score is 103 points

SECONDARY OUTCOMES:
Dermatology life quality index (DLQI) | Change from Baseline at 6th week and at 12th weeks of treatment
  DLQI consists of ten questions describe symptoms, feelings, leisure activities, work or school activities, personal relationships and treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Zizi Mohammed Ibrahim Ali, Riyadh, Saudi Arabia